

# The University of Alabama at Birmingham

# LAS CALLAHAN EYE

Department of Ophthalmology & Visual Sciences

July 7, 2025

# Manual of Procedures

Title of Project: Alabama Screening and Intervention for Glaucoma and Eye
Health through Telemedicine (AL-SIGHT)
Project dates: 9/30/2019 – 9/29/2024

Funding Agency: Centers for Disease Control and Prevention (1U01DP006441)

Date of this Document: June 18, 2025

Principal Investigators:

9/30/2019 – 4/30/2023: Lindsay A. Rhodes MD (contact PI), Christopher A. Girkin MD (PI)

5/1/2023 – 9/29/2024: Christopher A. Girkin MD (contact PI) 9/30/2024 – 7/1/2025: Cynthia Owsley PhD (contact PI)

### **Investigative Team:**

Lindsay A. Rhodes MD, Christopher A. Girkin MD, Cynthia Owsley PhD, Gerald McGwin Jr. PhD, Massimo Fazio PhD, Irfan M. Asif MD, Shilpa Register OD, Van Thi Ha Nghiem PhD, Ellen K. Antwi-Adjel OD, Thomas Swain PhD

### Clinical Research Staff Resources:

Angela McCombs BS (pre-award), Dylan McDonald MBA and Jennifer America MBM (post-award), Karen Searcey MSPH (regulatory), Mark Clark M.Eng (imaging manager), Liyan Gao PhD (Database designer/manager), Mitzi Swift BS, COT and Tara Sloan COT (clinical coordinators)

### **Table of Contents**

| | Page # |
|------------------------------|--------|
| 1. Aims of the Study | 3 |
| 2. Background | 4 |
| 3. Protocol | 9 |
| 4. Statistical Analysis Plan | 13 |
| 5. References | 14 |
| 6. Data Collection Forms | 20 |

### 1. Aims of the Study

Aim 1: Implement and evaluate a remote optic nerve assessment (RONA) protocol using telemedicine to identify glaucoma-associated disease in at-risk rural patients using portable multimodal structural and functional assessment of the optic nerve and retina. Also assess for diabetic retinopathy, cataract, visual acuity impairment, and refractive error.

Aim 2: Identify and evaluate remediation strategies for the barriers to patient adherence with referral and follow-up appointments by comparing the effectiveness of financial incentives along with a validated patient education program versus a validated patient education program alone.

Aim 3: Investigate the cost-effectiveness of the telemedicine program in diagnosing glaucoma using RONA versus usual in-person care from a glaucoma specialist.

### 2. Background

Prioritizing Vision Health. Vision health is an important public health concern affecting Americans of all ages. The 2016 report from the National Academies of Sciences, Engineering, and Medicine (NASEM) elevated the importance of a population health action framework that would transform "vision impairments from common to rare and eliminate correctable and avoidable vision impairments in the U.S. by 2030". The report also called on the Centers for Disease Control and Prevention (CDC) to develop a research agenda to provide evidence on effective policies, practices, and interventions that could delay the onset and progression of eye diseases and "achieve eye and vision health equity by improving care in underserved populations". Improving the "visual health of the nation through prevention, early detection, treatment, and rehabilitation" is also a Healthy People 2020 goal.<sup>3</sup> Specifically, this research plan focuses on a novel telemedicine-based care delivery model for the detection and management of the eye diseases of glaucoma, primarily, as well as other eye diseases such as diabetic retinopathy (DR). The public health challenge is that if eye conditions such as glaucoma and DR had been detected early in the disease course, vision impairment would be preventable, and sometimes reversible, with currently available ophthalmic treatments.

Epidemiology of Glaucoma. Glaucoma is one of the most common eye diseases of aging and is the leading cause of irreversible vision loss and blindness in older African Americans. Primary open angle glaucoma (POAG), the most common form of glaucoma, is a chronic progressive optic neuropathy traditionally characterized by changes in the optic disk, thinning of the retinal nerve fiber layer, and gradual loss of vision, with both peripheral vision and central vision affected depending on disease severity. The prevalence of POAG increases with age, affecting more than 1.8% of the population over 40 but increasing to 23.2% among African Americans and 9.4% among non-Hispanic whites over the age of 75.4 With the rapid growth in older populations, the number of POAG cases will increase 250% by 2050, directly affecting over 7 million lives. <sup>5</sup> These numbers are specifically for POAG and do not include those who are monitored and treated for elevated intraocular pressure or for glaucoma suspect status, which along with POAG can all be considered glaucoma associated diseases (GAD). While the number of patients with glaucoma will nearly double over the next 20 years, the number of US ophthalmologists is expected to grow only 0.67%.<sup>4,5</sup> The at-risk population for glaucoma in the U.S. is large, with older age as the primary risk factor as well as African Americans or Hispanics ≥ 40 years old, Asians, non-Hispanic whites ≥ 50 years old, older persons with diabetes, and those with a family history of glaucoma. POAG is at least 4-5 times higher in African Americans, progresses more rapidly and appears about 10 years earlier as compared to those of European descent. 6,7 Fortunately, vision loss from glaucoma can be prevented by early detection, consistent follow-up, and control of intraocular pressure with medication or surgery.

Epidemiology of Diabetic Retinopathy. Diabetes, and its ocular complications, is the leading cause of new cases of blindness in adults age 20-74 years in the US.<sup>8,9</sup> African Americans are 2 times more likely to have DR than whites. <sup>10</sup> In 2005-2008, 4.2 million (28.5%) Americans with diabetes ≥ age 40 had DR and of these, 655,000 (4.4%) had advanced DR that often leads to severe vision loss. 11 The number of people with DR is expected to increase more than 3-fold by 2050, creating an immense, costly public health problem. 9,12-14 Despite the risk of vision loss, only 50-60% of people with diabetes follow the recommendation to receive an annual dilated eye exam and this is even less in low-income and minority populations. 15-17 Successful management of DR includes early diagnosis, tight glycemic and blood pressure control, and medical or surgical treatment to prevent vision loss. 18-20

Epidemiology of Cataract and Refractive Error. Cataracts are a major cause of preventable visual impairment and blindness, especially in African Americans, with over 24 million people in the US having cataracts. 10 A major risk factor for cataracts is aging and thus there is an expected 50% increase in cataracts by 2030.<sup>21</sup> Additionally, studies have shown that African Americans have a reduced likelihood for curative cataract surgery, highlighting possible racial disparities in access to care for a reversible cause of visual impairment.<sup>22,23</sup> Refractive error is another major cause of preventable visual impairment in the US. Over 48 million people over age 40 in the US have refractive error, with the majority having myopia. Uncorrected refractive error has also been found to be associated with racial disparities.<sup>24</sup>

Personal Burden of Eye Disease. The personal burden of eye disease and its accompanying visual impairment is undisputed and widely documented. Adults with glaucoma experience reductions in health-related quality of life and mobility problems including ambulatory and driving difficulties and limitations in physical activity.<sup>25-41</sup> Persons with vision impairment, regardless of etiology, are at increased risk for depression, social disengagement, employment challenges, and problems accessing health care. 40,42-45 Several studies have demonstrated an association between vision impairment in adults and increased mortality risk, including studies focused on persons with glaucoma, cataract, and refractive error. 46-52 Thus, interventions to improve early detection, effective follow-up and implementation of evidence-based treatments for glaucoma, and patients' adherence to medication plans will improve the health and well-being of persons with this condition and at-risk for the condition.

Economic Burden of Eye Disease. The economic burden of eye disease in the U.S. is staggering. Analyses commissioned by the Centers for Disease Control and Prevention and Prevent Blindness America estimate the annual cost of adult vision problems in the U.S. at about \$139 billion.<sup>53</sup> In Alabama, the cost of vision problems is \$2.2 billion.<sup>53</sup> This includes U.S. economic factors such as direct medical costs, other direct costs (e.g., nursing home care stemming from vision impairment), and productivity losses (i.e., lower wages for Source: Rhodes LA, Girkin CA, Owsley C. Manual of Procedures, Alabama Screening and Intervention for 5 Glaucoma and Eye Health through Telemedicine (AL-SIGHT), Funded by Centers for Disease Control and

Prevention (1U01DP006441), Department of Ophthalmology & Visual Sciences, University of Alabama at

Birmingham, Heersink School of Medicine, 2024, Version 1.0.

visually impaired), as well as the financial burden incurred by the individual, caregivers, and other healthcare payers. The direct medical costs of glaucoma are \$5.8 billion/year, which does not include indirect costs such as incremental nursing home placements and productivity losses. For people aged 40- 64 years, the annual medical costs of glaucoma are \$1490/person and for those aged  $\geq$  65 years, they are \$2580/person. The annual medical costs of blindness and low vision per person from all causes, including glaucoma, are \$5870 and \$10,020 for people aged 40-64 years and  $\geq$  65 years, respectively. Costeffective benefits to quality of life have been reported for early detection and treatment of eye conditions such as glaucoma. Given projected Medicare shortfalls and potential reductions in Medicaid coverage, developing high quality and efficient means to provide care for these individuals will become increasingly important.

Barriers to Eye Care. Inadequate access to eye care delays diagnosis and increases the personal and economic burdens of eye disease and visual disability. For Problems accessing eye care are the most commonly cited barrier to care by African Americans in Alabama and elsewhere. For Sport Older African Americans are less likely to receive routine comprehensive eye care, when damaging eye conditions could be detected and treated early, and less likely to adhere to prescribed glaucoma therapies, thus contributing to higher rates of eye disease. The lower rate of receiving routine eye care may be contributing to higher rates of disability from eye disease. Factors underlying lower utilization include inadequate knowledge of basic symptoms, risk factors and available treatments; reduced financial resources; limited transportation; low trust in health care providers; and high cost. Tophthalmologists rarely practice in rural areas where African Americans represent the majority of the population in Alabama. This produces a problem accessing ophthalmological care, especially subspecialist care.

Alabama's Black Belt Region, named for its rich black soil, is a rural area with one of the highest poverty rates in the US. The Birmingham News has characterized it as America's Third World.<sup>67</sup> It has one of the highest concentrations of African American residents of any region of the country, representing over 50% of the population. In addition to having widespread poverty, the region is characterized by inadequate education, transportation, community resources, and a shortage of healthcare providers including a shortage of ophthalmologists and optometrists.<sup>66</sup>

To summarize, glaucoma is a blinding eye disease and a leading cause of irreversible vision loss in Americans, and THE leading cause in African Americans. In many rural counties in Alabama and the rest of the South, the majority of the population is African American. African Americans are less likely to receive routine, dilated comprehensive eye care that would facilitate early detection and thus prognosis. The number of cases of glaucoma and DR are expected to increase in the US. The personal burden of glaucoma, DR, cataract, refractive error, and vision impairment is heavy, with numerous negative implications for quality of life, and the economic burden is dramatically large. Ophthalmologists

specializing in glaucoma and retina are centered in urban areas, particularly in and around academic medical centers. Thus, all the factors we have discussed above -- the shortage of ophthalmologists in general but especially in communities with high concentrations of African Americans, the rising cost of care, and rapid growth in glaucoma prevalence in the population -- clearly necessitates an alternative model of care for these individuals.

Given the barriers to implementation of population-based screening for glaucoma, telemedicine is a potential strategy to improve disease detection and management as well as to improve effectiveness, access, and adherence with routine eye care. Telemedicine refers to the electronic communication of medical information from one site to another to improve a patient's clinical health status. 68 It has already been utilized in many healthcare fields and can improve health outcomes, increase accessibility to specialty care, and increase patient satisfaction.<sup>68,69</sup> By utilizing current technologies, telemedicine transmits patient data from a primary care clinic to another remote site for review by specialist physicians and thus, the standards of specialty care are more accessible to patients who live where no specialists practice. Telemedicine is well suited for the detection and management of certain eye conditions since there have been great strides made in the development of non-invasive ocular imaging devices that provide high levels of diagnostic reliability, ease of training of testing personnel, and electronically transmissible results. Telemedicine has been implemented in some areas of eye care but the vast majority of the literature on telemedicine for the chronic eye conditions of adulthood is focused on DR screening. Acceptance of telemedicine for DR using digital fundus photography has increased steadily around the world over the years stemming from its proven efficacy, costeffectiveness, and ability to reach underserved populations. 70-72

Applying Previous Experience in a New Way. This project focuses on the development and implementation of a community-based detection model for the two most common vision-threatening eye diseases in the African American population, POAG and DR. This will be achieved through a novel telemedicine program using RONA, based on integrated and collaborative partnerships, to improve both the quality of and access to eye care. The program will use advanced eye imaging technology to remotely assist in the detection and management of POAG, DR, cataract, and refractive error in a predominantly African American community receiving primary care through FQHC's in rural counties of Alabama, where African Americans represent 56% of the population. <sup>73</sup> Many of these rural counties are in Alabama's Black Belt Region that was described in detail above. Compared to many other states, Alabamians, particularly African Americans, have a disproportionately high prevalence of many risk factors for POAG and DR. Alabama has a higher prevalence of diabetes than any other state (~13%), and African American Alabamians have a diabetes mortality rate 2.5 times greater than white Alabamians.74 The relative lack of specialists in communities with high concentrations of African Americans, combined with the rapid growth in glaucoma and diabetes prevalence, clearly necessitates an innovative and community-based approach to eye care.

Achieving high levels of adherence to recommended health interventions has long been a challenge, particularly in rural, underserved populations. One method to try to increase adherence levels has been through financial incentives. Previous research in rural populations with improving adherence to preventive services such as mammography and influenza vaccination has shown that financial incentives are the only method to increase adherence compared to other behavioral interventions. 75 In addition to showing effectiveness of financial incentives, there are ethical considerations as to the appropriateness of incentivizing health behaviors through financial means. Shea et al. found that patients were willing to engage in incentive programs and had a positive experience without impact on the relationship with their physician. <sup>76</sup> In relation to eye care, Tan et al. found improved adherence to tertiary eye care services after community-based screenings in low socio-economic areas with the addition of an incentive care scheme.<sup>77</sup> That study provided a one-time transportation allowance to the appointment and a subsidy for the first tertiary eye care consultation.<sup>77</sup> In our proposed study, in addition to providing the eye health education program, financial incentives will also be used in the study sites in order to encourage patient adherence to referral and follow-up appointments.

### 2. Protocol

**Source Population**. This consisted of patients seeking healthcare at three FQHCs in north central Alabama. The three FQHCs are part of the Cahaba Medical Care Foundation, an Alabama-based FQHC. They care for a population of approximately 16,000 patients per year, including 58% who are African American, 38% White, and < 3% Hispanic. Among the active patients in these FQHCs, health insurance status is 25% Medicaid, 30% Medicare, 25% private insurance, and 20% uninsured. The study clinics are in rural Alabama towns: Centreville (Bibb County), Maplesville (Chilton County), and Marion (Perry County). This region of Alabama borders or is part of the region known as the Black Belt named for its rich black soil that supported cotton agriculture. In the 19th century, the agricultural workers were enslaved African Americans. The Black Belt consists of 9 of 10 of the poorest counties in the state. Poverty is directly link to health disparities in the Black Belt. Today this region's population is over 50% African American.

**Inclusion criteria.** Patients presenting at these clinics were eligible to participate if they had one or more risk factors for  $GAD^{79}$  and volunteered to participate: (1) African American or His-panic  $\geq$ 40 years of age; (2) White  $\geq$ 50 years of age; (3) anyone  $\geq$ 18 years of age with diabetes, (4) anyone  $\geq$ 18 years of age with a GAD; and (5) anyone  $\geq$ 18 years of age with a family history of glaucoma. All participants spoke and understood English.

**Exclusion criterion:** If patients did not complete written informed consent to participate, they did not participate.

Study Design. This study had two arms. The protocol, as described below, was identical in both arms, except for the following. One arm consisted of participants not receiving any financial incentive for attending recommended follow-up care with an optometrist or ophthalmologist based on positive eye screening results. The other arm had a financial incentive, that is, participants recommended to attend a follow-up care exam with an optometrist or ophthalmologist received \$50 for attending the appointment. In the second arm, we confirmed with the eye care provider through the optometrist's or ophthalmologist's electronic medical records (EMR) whether the participant attended the follow-up appointment. We considered randomizing patients to each of the two arms. We decided not to use this approach because we were concerned that patients may talk among themselves (they live in small rural communities) about some receiving a financial incentive to attend recommended follow-up visits versus others not receiving a financial incentive. This was viewed as causing a potential conflict for patients in terms of their participating in the study and viewed as potentially unfair by patients. Thus, our approach was to first enroll half of the total number of patients in the non-financial incentive arm, and then when that was complete, to enroll the second half of the total number of patients in the financial arm. The goal was to enroll 500 patients in each arm.

**Protocol Measurements**. These are each described below. All were completed in a single visit to the FQHC. All eye and visual function measurements were performed on each eye separately. The clinical coordinators (certified ophthalmic technicians) collected all data including questionnaires.

**Demographic review.** Questionnaires obtained information on birthdate, gender, race, ethnicity, marital status, medical insurance status, transportation availability, education level, employment status, whether they received an eye examination in the past two years, reasons for not seeking an eye examination in the past two years, and contact information (address, phone number).

**Self-reported clinical characteristics**. Questionnaires obtained information on the following: smoking status, family history of glaucoma or blindness, and ocular history of major chronic eye diseases or conditions. Family history of glaucoma was considered positive if a participant reported a glaucoma diagnosis for a first degree relative (parent, sibling, child).

Ocular screening. All measurements were completed under undilated conditions, as follows. (1) Distance visual acuity was assessed using a Snellen chart presented at 20 feet while participants wore whatever correction (if any) they were habitually wearing for distance. (2) Autorefraction was carried out with the QuickSee (PlenOptika Inc) or Retinomax (Nikon). (3) Intraocular pressure (IOP) was measured with the iCare portable rebound tonometer (iCare USA). A second measurement was taken if the IOP was > 21 mm Hg. If these 2 IOPs differed by more than 2 mm Hg, a third measurement was taken. If IOP was measured twice, the mean value was used as the IOP; if it was measured 3 times, the middle value was used. Participants with IOP ≥ 30 mm Hg were referred to an optometrist or ophthalmologist in our fast-track protocol: IOP > 30 mm Hg within 2 weeks; IOP > 35 mm Hg, within 1 week; and IOP > 40 mm Hg, an urgent referral within 1 day. (4) Visual field was assessed using three methods: the Humphrey Field Analyzer 3 (HFA3) using the Swedish Interactive Threshold Algorithm Fast screening strategy (Carl Zeiss Meditec), the Melbourne Rapid Fields, a tablet-based perimetry test (M&S Technologies), and the Alleye test (Oculocare Medical).

**Retinal imaging.** Spectral domain optical coherence tomography (SD- OCT) was performed using the Maestro2 (Topcon Medical Systems), measuring the thickness of the retinal nerve fiber layer of the optic nerve head and of the macula by a single widefield OCT scan measuring 12 ×9 mm (512 ×128 pixels). This encompassed both the macula and disc. The Maestro2 also provided high-resolution fundus photographs encompassing both the optic nerve and macula.

**Telemedicine.** All the above ocular screening data and retinal imaging, as well as the medical and ocular history and demographics (age, gender, race, ethnicity) were

electronically transferred to a remotely located glaucoma-fellowship-trained ophthalmologist for reading and interpretation. With respect to visual field data, only HFA3 data were transferred since the other two field tests are not routinely used in standard of care in glaucoma assessments. The ophthalmologist made the following diagnostic judgments based on the screening in terms of the presence of the following conditions: glaucoma, glaucoma suspect, ocular hypertension, diabetic retinopathy, cataract, refractive error, or any other ocular conditions identified through the above screening data.

Diagnoses for GAD conditions are as follows. Ocular hypertension is defined as no glaucomatous appearing disc changes (described below), a normal visual field (described below), and statistically elevated IOP ≥23 mm Hg. Glaucoma suspect is defined as the presence of glaucomatous-appearing disc changes (de-scribed below), normal visual field (described below), and statistically normal IOP < 23 mm Hg. Glaucoma refers to the presence of glaucomatous appearing disc changes (de-scribed below) and an abnormal visual field (described be-low). A glaucomatous appearing optic disk is defined as evidence of excavation, neuroretinal rim thinning or notching, localized or diffuse retinal nerve fiber layer (RNFL) defect, or a between-eye asymmetry of the vertical cup disc ratio > 0.2. A glaucomatous visual field defect is defined as a reliable SAP Humphrey 24-2 field (defined as < 33% false-positives results, false-negative results, and fixation losses) that exhibits a pattern standard deviation outside of the 95% normal limits, or a glaucoma hemifield test outside of the 99% normal limits consistent with an RNFL defect pattern based on clinical review. A normal eye that meets none of these definitions of GAD is defined as not having glaucomatous-appearing disc changes and having a normal visual field and statistically normal IOP < 23 mm Hg (both described above). Diagnoses of DR were made based on the National Health Service Grading Classification System.80

Each participant, the FQHC primary care provider, and their eye care provider (if they had one) received the final report about the ophthalmologist's screening-based diagnoses. These were sent out electronically within 14 days of the participant's screening visit date. The report contained diagnostic information on the conditions mentioned above plus visual acuity, IOP, recommended treatment, and whether a follow-up exam was recommended.

Recommendations from the telemedicine ophthalmologist. Participants whom the ophthalmologist clinically judged as normal were recommended to undergo an annual comprehensive eye examination on a routine basis. The following participants were recommended for a follow-up examination visit with an optometrist who was partnered with the FQHC (located in a separate office), or an ophthalmologist at the Glaucoma Service at UAB, the Lions Eye Clinic at UAB, or an ophthalmologist whose clinic was located in the FQHC geographic area: participants with 20/40 or worse visual acuity and/or with an IOP ≥23 mm Hg in either eye, as well as those with GAD (glaucoma, glaucoma suspect, or ocular hypertension), DR, and/or other ocular condition that the ophthalmologist viewed as needing to be examined in per- son. The FQHC staff scheduled

the appointment and communicated the details to the participant. The study coordinator followed up with the clinic where participants were scheduled for the follow-up examination to determine whether they actually attended the appointment by contacting the eye clinic and getting confirmation through the EMR.

Vision-Specific Health-Related Quality of Life. This was assessed using the National Eye Institute Visual Function Question – 9.81

Satisfaction with the RONA screening. Following the ocular screening, participants' satisfaction with the telemedicine screening was evaluated by a questionnaire using Likert scales. Questions address satisfaction with the vision screening and the time that it took to complete it (very satisfied/satisfied/dissatisfied/very dissatisfied), as well as how convenient the venue was (very convenient/convenient/inconvenient/very inconvenient). Participants were also asked whether they would recommend the ocular screening to others, whether they could return to the same venue in 12 months for another screening, and whether they could make a follow-up visit to an optometrist or ophthalmologist if referred for a problem identified by the screening (very likely/somewhat likely/not very likely/not at all likely)

### 4. Statistical Analysis Plan

Demographic, socioeconomic, medical, and ocular factors were compared across groups who did and did not receive incentives for obtaining follow-up care using unpaired t-tests for continuous data and using the Fisher's exact test for categorical data. The proportion of individuals in each group who were recommended for a follow-up comprehensive eye exam and, among those individuals, the proportion who attended that exam was compared using chi-square tests. Given the demographic differences in the study groups, the impact of incentivization was evaluated using a subset of incentivized and non-incentivized patients matched on age, sex and race. The impact of COVID-19 on follow-up attendance was estimated by correlating the rate of COVID-19 deaths in Alabama obtained from the Alabama Department of Public Health and the average number of daily hospitalizations per month with the proportion of those attending follow-up referrals during each month of the study. P-values ≤ 0.05 (two-sided) were considered statistically significant.

### 5. References

- 1. Teutsch SM, McCoy MA, Woodbury RB, Welp A. Making eye health a population health imperative: Vision for tomorrow. Washington DC: The National Academies Press;2016.
- Todd J, Whitson HE, Marshall EC. Eye and vision health for tomorrow: Recommendations to coordinated action. JAMA Ophthalmology. 2019;137(2):208-211.
- 3. National Center for Health Statistics. Healthy People 2020 <a href="https://www.cdc.gov/nchs/healthy\_people/hp2020.htm">https://www.cdc.gov/nchs/healthy\_people/hp2020.htm</a>. Centers for Disease Control and Prevention 2020.
- 4. Friedman DS, Wolfs RC, O'Colmain BJ, Klein BE, Taylor HR, West S, Leske MC, Mitchell P, Congdon N, Kempen J. Prevalence of open-angle glaucoma among adults in the United States. Archives of Ophthalmology. 2004;122:532-538.
- 5. Vajaranant TS, Wu S, Torres M, Varma R. The changing face of primary open-angle glacuoma in the United States: demographics and geographic changes from 2011 to 2050. American Journal of Ophthalmology. 2012;154(2):303-314.
- 6. Lafuma AJ, Brezin AP, Fagnani FL, Mesbah M, Berdeaux GH. Prevalence of visual impairment in relation to the number of ophthalmologists in a given area: a nationwide approach. Health and Quality of Life Outcomes. 2006;4:34.
- 7. Javitt JC, Bean AM, Nicolson GA, Babish JD, Warren JL, Krakauer H. Undertreatment of glaucoma among black Americans. New England Journal of Medicine. 1991;325:1418-1422.
- 8. Congdon N, O'Colmain B, Klaver CC, Klein R, Munoz B, Friedman DS, Kempen J, Taylor HR, Mitchell P. Causes and prevalence of visual impairment among adults in the United States. Archives of Ophthalmology. 2004;122:477-485.
- 9. Lee PP, Feldman ZW, Osterman J, Brown DS, Sloan FA. Longitudinal prevalence of major eye diseases. Archives of Ophthalmology. 2003;121:1303-1310.
- 10. Sommer A, Tielsch JM, Katz J, Quigley HA, Gottsch JD, Javitt JC, Martone JF, Royall RM, Witt KA, Ezrine S. Racial differences in the cause-specific prevalence of blindness in east Baltimore. The New England Journal of Medicine. 1991;325(20):1412-1417.
- 11. Centers for Disease Control and Prevention. National diabetes fact sheet: National estimates and general information on diabetes and prediabetes in the United States, 2011. Atlanta, GA: US Department of Health and Human Services.;2011.
- 12. Vitale S, Cotch MF, Sperduto RD. Prevalence of visual impairment in the United States. JAMA. 2006;295:2158-2163.
- 13. Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF, Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Archives of Ophthalmology. 2004;122(4):552-563.

- 14. Saaddine JB, Honeycutt AA, Narayan KM, Zhang X, Klein R, Boyle JP. Projection of diabetic retinopathy and other major eye diseaes among people with diabetes mellitus: Unisted States, 2005-2050. Archives of Ophthalmology. 2008;126:1740-1747.
- 15. Zhang X, Saaddine J, Lee P, Grabsowski D, Kanjilal S, Duenas M, Narayan K. Eye Care in the United States...Do we deliver to high risk people who can benefit most from it? Archives of Ophthalmology. 2007;125:411-418.
- 16. Schoenfeld ER, Greene JM, Wu SY, Leske C. Patterns of adherence to diabetes vision care guidelines. Ophthalmology. 2001;108:563-571.
- 17. MacLennan PA, McGwin GJ, Heckemeyer C, Lolley VR, Hullett S, Saaddine J, Shrestha S, Owsley C. Eye care utilization among a high-risk diabetic population seen in a public hospital's clinics. JAMA Ophthalmology. 2014;132:162-167.
- 18. Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. Glycosylated hemoglobin predicts the incidence and progression of diabetic retinopathy. JAMA. 1988;260:2864-2871.
- 19. Rowe S, MacLean CH, Shekelle PG. Preventing visual loss from chronic eye disease in primary care. Journal of the American Medical Association. 2004;291:1487-1496.
- 20. Diabetic Retinopathy Study Research Group. Photocoagulation treatment of proliferative diabetic retinopathy: Clinical application of diabetic retinopathy study (DRS) findings, DRS report number 8. Ophthalmology. 1981;88:583-600.
- 21. National Eye Institute (NIH) Cataracts. <a href="http://www.nei.nih.gov/eyedata/cataract.asp#3b">http://www.nei.nih.gov/eyedata/cataract.asp#3b</a>. Accessed February 1, 2019.
- 22. Kauh cY, Blachley TS, Lichter PR, Lee PP, Stein JD. Geographic variation in the rate and timeing of cataract surgery among US communities. JAMA Ophthalmology. 2016;134(3):267-276.
- 23. Javitt JC, Kendix M, Tielsch JM, Steinwachs DM, Schein OD, Kolb MM, Steinberg EP. Geographic variation in utilization of cataract surgery. Medical Care. 1995;33(1):90-105.
- 24. Qiu M, Wang SY, Singh K, Lin SC. Racial disparities in uncorrected and undercorrected refractive error in the United States. Investigative Ophthalmology & Visual Science. 2014;55(10):6996-7005.
- 25. Wilson MR, Coleman AL, Yu F, Bing EG, Sasaki IF, Berlin K, Winters J, Lai A. Functional status and well-being in patients with glaucoma as measured by the medical outcomes study short form-36 questionnaire. Ophthalmology. 1998;105:2112-2116.
- 26. Gutierrez P, Wilson MR, Johnson C, Gordon M, Cioffi GA, Ritch R, Sherwood M, Meng K, Mangione CM. Influence of glaucomatous visual field loss on health-related quality of life. Archives of Ophthalmology. 1997;115:777-784.
- 27. Parrish RK, II, Gedde SJ, Scott IU, Feuer WJ, Schiffman JC, Mangione CM, Montenegro-Piniella A. Visual function and quality of life among patients with glaucoma. Archives of Ophthalmology. 1997;115:1447-1455.

- 28. Sherwood MB, Garcia-Siekavizza A, Meltzer MI, Hebert A, Burns AF, McGorray S. Glaucoma's impact on quality of life and its relation to clinical indicators: A pilot study. Ophthalmology. 1998;105:561-566.
- 29. Janz NK, Wren PA, Lichter PR, Musch DC, Gillespie BW, Guire KE, Group TCIGTS. Quality of life in newly diagnosed glaucoma patients: The collaborative initial glaucoma treatment study. Ophthalmology. 2001;108:887-898.
- 30. Aspinall PA, Hill AR, Nelson P, O'Brien C, O'Connell E, McCloughan L, Azuara-Blanco R, Brice R, Green S, Steeds C. Quality of life in patients with glaucoma: A conjoint analysis approach. Vision Impairment Research. 2005;7:13-26.
- 31. Spaeth G, Walt J, Keener J. Evaluation of quality of life for patients with glaucoma. American Journal of Ophthalmology. 2006;141:S3-S14.
- 32. Ringsdorf L, McGwin GJ, Owsley C. Visual field defects and vision-specific health-related quality of life in African Americans and whites with glaucoma. Journal of Glaucoma. 2006;15:414-418.
- 33. McGwin GJ, Xie A, Mays A, Joiner W, DeCarlo DK, Hall TA, Owsley C. Visual field defects and the risk of motor vehicle collisions among patients with glaucoma. Investigative Ophthalmology and Visual Science. 2005;46:4437-4441.
- 34. Haymes SA, LeBlanc RP, Nicolela MT, Chiasson LA, Chauhan BC. Risk of falls and motor vehicle collisions in glaucoma. Investigative Ophthalmology and Visual Science. 2007;48:1149-1155.
- 35. Haymes S, LeBlanc R, Nicolela M, Chiasson L, Chauhan B. Glaucoma and on-road driving performance. Investigative Ophthalmology & Visual Science. 2008;49(7):3035-3041.
- 36. Turano KA, Rubin GS, Quigley HA. Mobility performance in glaucoma. Investigative Ophthalmology and Visual Science. 1999;40(12):2803-2809.
- 37. Geruschat D, Turano K. Estimating the amount of mental effort required for independent mobility: persons with glaucoma. IOVS. 2007;48(9):3988-3994.
- 38. Bowers A, Peli E, Elgin J, McGwin G, Owsley C. On-road driving with moderate visual field loss. Optometry and Vision Science. 2005;82(8):657-667.
- 39. Ramulu PY, Hochberg C, Maul EA, Chan ES, Ferrucci L, Friedman DS. Glaucomatous visual field loss associated with less travel from home. Optometry and Vision Science. 2014;91:187-193.
- 40. Curriero FC, Pinchoff J, van Landingham SW, Ferrucci L, Friedman DS, Ramulu PY. Alternation of travel patterns with vision loss from glaucoma and macular degeneration. JAMA Ophthalmology. 2013;131:1420-1426.
- 41. Black AA, Wood JM, Lovie-Kitchin JE. Inferior field loss increases rate of falls in older adults with glaucoma. Optometry and Vision Science. 2011;88:1275-1282.
- 42. Black AA, Wood JM, Lovie-Kitchin JE. Inferior visual field reductions are associated with poorer functional status among older adults with glaucoma. Ophthalmic Physiological Optics. 2011;31:283-291.
- 43. Crudden A, McBroom L. Barriers to employment: a survey of employed persons who are visually impaired. Journal of Visual Impairment & Blindness. 1999;93:341-350.

- 44. Rees G, Tee HW, Marella M, Fenwick E, Dirani M, Lamoureux EL. Vision-specific distress and depressive symptoms in people with vision impairment. Investigative Ophthalmology and Visual Science. 2010;51(6):2891-2896.
- 45. Jones G, Rovner B, Crews J, Danielson M. Effects of depressive symptoms on health behavior practices among older adults with vision loss. Rehabilitation Psychology. 2009;54(2):164-172.
- 46. Zheng DD, Christ SL, Lam BL, Arheart KL, Galor A, Lee DJ. Increased mortality risk among the visual impaired: The roles of mental well-being and preventive care practices. Investigative Ophthalmology & Visual Science. 2012;53:2685-2692.
- 47. McCarty CA, Nanjan MB, Taylor HR. Vision impairment predicts 5 year mortality. British Journal of Ophthalmology. 2001;85:322-326.
- Lee DJ, Gomez-Marin O, Lam BL, Zheng DD. Visual acuity impairment and mortality 48. in US adults. Archives of Ophthalmology. 2002;120:1544-1550.
- 49. Knudtson MD, Klein BE, Klein R. Age-related eye disease, vision impairment, and survival: the Beaver Dam Eye Study. Archives of Ophthalmology. 2006;124:243-249.
- 50. Egge K, Zahl PH. Survival of glaucoma patients. Acta Ophthalmologica Scandinavia. 1999;77:397-401.
- Lee DJ, Gomez-Marin O, Lam BL, Zheng DD. Glaucoma and survival: the National 51. Health Interview Survey 1986-1994. Ophthalmology. 2003;110:1476-1483.
- 52. Owsley C, McGwin G, Jr., Scilley K, Meek GC, Seker D, Dyer A. Effect of refractive error correction on health-related quality of life and depression in older nursing home residents. Archives of Ophthalmology. 2007;125(11):1471-1477.
- 53. Wittenborn JS, Rein DB. Cost of vision problems: the economic burden of vision loss and eye disorders in the United States. Prevent Blindness America, Chicago IL: NORC at the University of Chicago; 2013.
- 54. Leske MC, Heijl A, Hussein M, Bengtsson B, Hyman L, Komaroff E, Early Manifest Glaucoma Trial Group. Factors for glaucoma progression and the effect of treatment: the early manifest glaucoma trial. Archives of Ophthalmology. 2003;121:48-56.
- 55. Rein DB, Wittenborn BS, Lee, PP, Wirth KE, Sorensen SW, Hoerger TJ, Saaddine JB. The cost-effectiveness of routine office-based identification and subsequent medical treatment of primary open-angle glaucoma in the United States. Ophthalmology. 2009;116:823-832.
- 56. Prevent Blindness America and National Eye Institute. Vision problems in the U.S.: Prevalence of adult vision impairment and age-related eye disease in America. 2002.
- Owsley C, McGwin G, Scilley K, Girkin CA, Phillips JM, Searcey K. Perceived barriers 57. to care and attitudes about vision and eye care: Focus groups with older African Americans and eye care providers. Investigative Ophthalmology and Visual Science. 2006;47(7):2797-2802.

- 58. Owsley C, McGwin GJ, Weston J, Stalvey BT, Searcey K, Girkin CA. Preliminary evaluation of the InCHARGE program among older African Americans in rural Alabama. Journal of Health Disparities Research and Practice. 2010;3:115-126.
- 59. Centers for Disease Control and Prevention. Reasons for not seeking eye care among adults aged ≥ 40 years with moderate-to-severe visual impairment -- 21 states, 2006-2009. Morbidity Mortality Weekly Report. 2011;60:610-613.
- 60. Tielsch JM, Sommer A, Katz J, Royall RM, Quigley HA, Javitt JC. Racial variations in the prevalence of primary open-angle glaucoma. JAMA. 1991;266:369-374.
- 61. Bazargan M, Baker RS, Bazargan S. Correlates of recency of eye examination among elderly African-Americans. Ophthalmic Epidemiology. 1998;5(2):91-100.
- 62. Wang F, Javitt J, Tielsch J. Racial variations in treatment for glaucoma and cataract among medicare recipients. Ophthalmic Epidemiology. 1997;4(2):89-100.
- 63. Dreer LE, Girkin C, Mansberger SL. Determinants of medication adherence to topical glaucoma therapy. Journal of Glaucoma. 2012;21(4):234-240.
- 64. Walker EA, Basch CE, Howard CJ, Zybert PA, Kromholz WN, Shamoon H. Incentives and barriers to retinopathy screening among African-Americans with diabetes. Journal of Diabetes Complications. 1997;11:298-306.
- 65. Ellish N, Royak-Schaler R, Passmore S, Higginbotham E. Knowledge, attitudes, and beliefs about dilated eye examinations among African-Americans. Investigative Ophthalmology & Visual Science. 2007;48(5):1989-1994.
- 66. MacLennan PA, Owsley C, Searcey K, McGwin GJ. A survey of Alabama eye care providers in 2010. BMC Ophthalmology. 2014;3:44.
- 67. BirminghamNews. Special Report. The Black Belt. Alabama's Third World. Birmingham AL2002.
- 68. American Telemedicine Association. What is telemedicine?

  <a href="http://www.americantelemed.org/about-telemedicine/what-is-telemedicine#.VNUTSSmJf\_A">http://www.americantelemed.org/about-telemedicine/what-is-telemedicine#.VNUTSSmJf\_A</a>. Published 2014. AccessedAugust 2, 2024.
- 69. Rhodes LA, Huisingh CE, McGwin GJ, Mennemeyer ST, Bregantini M, Patel N, Wiley DM, LaRussa R, Box D, Saaddine J, Crews JE, Girkin CA, Owsley C. Eye care quality and accessibility improvement in the community (EQUALITY): impact of an eye health education program on patient knowledge about glaucoma and attitudes about eye care. Patient Related Outcome Measures. 2016;7:37-48.
- 70. Au A, Gupta O. The economics of telemedicine for vitreoretinal diseases. Current Opinion in Ophthalmology. 2011;22:194-198.
- 71. Murchison AP, Haller JA, Mayro EL, Hark LA, Gower EW, Huisingh C, Rhodes LA, Friedman DS, Lee DJ, Lam BL, Innovative Network for Sight (INSIGHT) Research Group. Reaching the unreachable: Novel approaches to telemedicine screening of underserved populations for vitreoretinal disease. Current Eye Research. 2017;42(7):963-970.
- 72. Kawaguchi A, Sharafeldin N, Sundarum A, Campbell S, Tennant M, Rudinsky C, Weis E, Damji KF. Tele-ophthalmology for age-related macular degeneration and diabetic

- retinopathy screening: A systematic review and meta-analysis. Telemedicine Journal and e-Health. 2018;24(4):301-308.
- 73. US Census Bureau. <a href="http://quickfacts.census.gov/qfd/states/01000.html">http://quickfacts.census.gov/qfd/states/01000.html</a>.
- Centers for Disease Control and Prevention. Compressed Mortality File, 199-2008. 74. http://wonder.cdc.gov/ucd-icd10.html: National Center for Health Statistics, Atlanta GA.
- 75. Shekelle P, Stone EM, Maglione M, Hirt M, Mojica W, Srikanthan P, Tomizawa T, Morton S, roth EA, Chao B, Breuder T, Jackson J, Rhodes SD, Mittman B, Grimshaw J, Rubenstein L, Reubenstein L. Interventons that increase the utilization of medicarefunded preventive services for persons age 65 and older. US Department of Health and Human Services, Health Care Financing Administration; 2004.
- 76. Shea JA, Adejare A, Volpp KG, Troxel AB, Finnerty D, Hoffer K, Isaac T, Rosenthal M, Seguist TD, Asch DA. Patients' views of a behavioral intervention including financial incentives. Americal Journal of Managed Care. 2017;23(6):366-371.
- 77. Tan AC, Man R, Wong CW, Lee SY, Lamoureux EL. Randomized controlled trial evaluating a novel community eye care programme for elderly individuals with visual impairment. Clinical & Experimental Ophthalmology. 2018;46(6):593-599.
- Aladuwaka S, Alagan R, Singh R, Mishra M. Health burdens and SES in Alabama: 78. Using geographic information system to examine prostate cancer health disparity Cancer. 2022;14(19):4824.
- 79. Stein JD, Khawaja AP, Weizer JS. Glaucoma in adults — screening, diagnosis, and management. JAMA. 2021;325(2):164-174.
- 80. Harding SP, Greenwood R, Adlington S, Gibson J, Owens DA, Talylor R, Kohner EM, Scanlon P, Leese G, Diabetic Retinopathy Grading and Disease Management Working Party. Grading and disease management in national screening for diabetic retinopathy in England and Wales. Diabetic Medicine. 2003;20:965-971.
- Kodjebacheva G, Coleman AL, Ensrud KE, Cauley JA, Yu F, Stone KL, Pedula KL, 81. Hochberg MC, Mangione CM. Reliability and validity of abbreviated surveys derived from the National Eye Institute Visual Function Questionnaire. American Journal of Ophthalmology. 2010;149:330-340.

# 6. Data Collection Forms Data collection forms are appended to this document.

## **Baseline Intake and Education Form**

| Record ID | | |
|---|---|---|
| START TIME Intake and Consent | | |
| Subject Name/Initials: | | |
| Study ID | {Study ID= CDC + Initials + Recor | d ID) |
| Date of Baseline Intake | , | |
| Form Completed By (Initials/#) | - | |
| ELIGIBILITY CRITERIA | | |
| What is Your Date of Birth?<br>(If born after 2002 participant is not eligible) | (MM-DD-YYYY) | |
| What is Your Age? | , | |
| Which Cahaba Medical Care Clinic do you see your primary care Centreville ( 405 Belcher Street, Centreville, AL 35042) Maplesville (9431 Alabama 22, Maplesville, AL 36750) Marion (1303 Washington Street, Marion, AL 36756) Woodstock (28921 Highway 5, Woodstock, AL 35188) West Blocton (319 Magnolia Street, West Blocton, AL 35184) Bessemer (975 9th AVE SW, Bessemer, AL 35022) | provider? | |
| CONFIRM ADDRESS FOR ELIGIBILITY AND MAILINGS | | |
| Mailing address street and apartment number | (address and apartment number) | |
| City, State, Zipcode | | |
| | (city, state and zip code) | |

03/20/2023 3:38pm

projectredcap.org



### Please ask subjects for phone numbers and email addresses so we can contact them after the eye screening with results and schedule a follow-up eye doctor appointment if needed. If you have a telephone, what is the number (cell or home)? ○ Yes ○ No ○ Not sure If you use text messaging on your cell phone, do you have an unlimited monthly plan? O Getting new plan, so yes If you use email, what is your email address? ☐ Phone call What are the best WAYS to reach you about your eye ☐ Mail health? ☐ Text Message ☐ Email What are the best TIMES OF THE DAY to reach you about ☐ Moming your vision health? ☐ Afternoon ☐ Evening Do you have a family member or caregiver that we can ○ Yes ○ No contact in case of an eye care emergency? Names and phone number(s) of family or a caregiver that we can contact and how they are related to you (son, daughter, sister)? What is your gender? Other O Prefer not to say Do you consider yourself of Hispanic, Latino or ○ Yes ○ No Spanish Origin? ○ African American/ Black ○ American Indian/ Alaska Native ○ Asian ○ Native Hawaiian or Paging How do you self-identify your race? Native Hawaiian or Pacific Islander White Multiracial Ounknown/ Not Reported/ Refused to answer What is your marital status? Do you have health insurance? ○Yes ○No

REDCap 03/20/2023 3:38pm projectredcap.org

| If yes, which type(s)? | |
|---|---|
| ☐ Private insurance ☐ Medicare ☐ Medicaid ☐ Supp | lemental insurance |
| Do you have any type of health insurance coverage for eye care or vision? | <ul><li>Yes</li><li>No</li><li>Not Sure</li></ul> |
| If our eye doctors recommend you need follow-up eye care, with you? | do you have a family, friend, or caregiver that could go |
| ○ Yes ○ No ○ Maybe, Not sure | |
| How did you travel to get here today? | ☐ Drove myself ☐ Another person drove me ☐ Bus or other public transportation ☐ Walked ☐ Rode a bike ☐ Taxi ☐ Other: |
| If other transportation today, please specify | · |
| If our eye doctors recommend you need follow-up eye care in Birmingham or Centreville, check all ways you may be able to travel there? | ☐ Drive myself ☐ Another person will drive me ☐ Bus or other public transportation ☐ Walk ☐ Ride a bike ☐ Taxi ☐ Other: |
| If other transportation for follow up, please specify | |
| Employment status: please choose 1 response Are you currently: | Employed full-time for wages Employed part-time for wages Self-employed Unemployed Retired Unable to work/disabled A caregiver/homemaker A student Other Prefer not to answer/don't know |
| Last level of education completed: | <ul> <li>Less than high school</li> <li>High school of equivalent</li> <li>Some college or associate's degree</li> <li>College graduate</li> <li>Graduate School</li> <li>PhD or other professional degree (MD, JD, etc)</li> <li>Prefer not to answer</li> </ul> |

REDCap\* 03/20/2023 3:38pm projectredcap.org

| Now I am going to ask you some questions about cost. | |
|---|---|
| Is the cost of an eye exam a problem for you? | <ul> <li>Not a problem at all</li> <li>A little bit of a problem</li> <li>Somewhat of a problem</li> <li>A big problem</li> </ul> |
| Is the cost of buying eyeglasses a problem for you? | Not a problem at all A little bit of a problem Somewhat of a problem A big problem |
| If the doctor prescribed eye drops for you in order to treat an eye problem you have, would the cost of prescription eye drops be a problem for you? | Not a problem at all A little bit of a problem Somewhat of a problem A big problem |
| EDUCATION Questions | |
| 1. It is important to go to the eye doctor at least once every two years. | <ul><li>○ Strongly agree</li><li>○ Somewhat agree</li><li>○ Somewhat disagree</li><li>○ Strongly disagree</li></ul> |
| 2. A person can have glaucoma and not know it. | <ul><li>○ True</li><li>○ False</li><li>○ Not sure</li></ul> |
| 3. Glaucoma can be controlled. | <ul><li>○ True</li><li>○ False</li><li>○ Not sure</li></ul> |
| 4. Vision loss from glaucoma can be restored. | <ul><li>○ True</li><li>○ False</li><li>○ Not sure</li></ul> |
| 5. A complete glaucoma exam consists only of measuring eye pressure. | <ul><li>○ True</li><li>○ False</li><li>○ Not sure</li></ul> |
| 6. People at risk for glaucoma should have an eye examination through dilated pupils. | <ul><li>○ True</li><li>○ False</li><li>○ Not sure</li></ul> |
| 7. There is no need to go to the eye doctor if you are not having a problem with your eyes. | <ul> <li>Strongly agree</li> <li>Somewhat agree</li> <li>Somewhat disagree</li> <li>Strongly disagree</li> </ul> |
| END TIME of Baseline Intake and Education | |
| Warning: It has been over 30 minutes since the start time. Please check the start time and end time on this form | ○ Yes ○ No<br>(The time period is over 30 minutes.) |

03/20/2023 3:38pm projectredcap.org **REDCap**°

# **Medical and Ocular History**

| Record ID | |
|---|---|
| START TIME Ocular and Medical History | |
| Subject Name/Initials: | |
| Study ID | |
| | (Study ID= CDC + Initials + Record ID) |
| Date Medical and Ocular History | |
| Medical and ocular history completed by | ○ UAB team ○ Self-Administered |
| Form completed by (Name/#) | |
| MEDICAL HISTORY | |
| Have you been diagnosed with any of the following medical | conditions? |
| None □ Diabetes □ High blood pressure □ Heart □ Asthma, COPD/emphysema □ Insomnia □ Cognitive □ Arthritis or osteoporosis □ Hearing problems □ Fool problems | impairment Depression |
| If you have diabetes, do you know your last A1C level? | ○ Yes ○ No |
| Diabetes (1=Yes, 0=No) | |
| If you have diabetes and know your last A1C level, what was your last A1C level? | |
| Do you currently smoke cigarettes? | ○ Yes ○ No |
| Have you ever smoked a pack a day for more than one | ○ Yes ○ No |

REDCap\* 03/20/2023 3:39pm projectredcap.org

| OCULAR HISTORY | |
|---|---|
| Have you ever had an eye exam? | ○ Yes ○ No |
| If you have seen an eye care provider, we would be happy t<br>provider. Would you like us to send your vision screening re | |
| ○ Yes ○ No | |
| Eye Care Provider<br>Name, Address<br>Telephone | |
| Do you wear prescription eye glasses? | ○ Yes ○ No |
| If YES, how old are your prescription eye glasses? | |
| O Less than 1 year O Less than 2 years O More than | 2 years O Can't remember |
| When was the last time you saw any eye care provider to ch | neck your vision and glasses prescription? |
| ○ This year ○ Within two years ○ More than 2 years | ○ Can't remember ○ Never had an eye exam |
| When was the last time you had an eye exam by any eye ca | are provider where your eyes were dilated? |
| ○ This year ○ Within two years ○ More than 2 years | ○ Can't remember ○ Never had an eye exam |
| What is the main reason you have not visited an eye care professional in the past 2 years? (1 response) | <ul> <li>Cost of eye exam</li> <li>Do not have vision insurance</li> <li>Do not have/know an eye doctor</li> <li>Cannot get to the office/clinic (too far away, no transportation)</li> <li>Could not get an appointment</li> <li>No reason to go (no problem)</li> <li>Have not thought of it</li> <li>Other</li> </ul> |
| Do you have any of the following eye conditions? | None Need Eye Glasses (Refractive error) Dry Eye Blurry Vision Double vision Cataract High Eye Pressure Glaucoma or Glaucoma Suspect Diabetic Retinopathy (diabetic eye disease) Macular Degeneration Floaters Narrow Angle Ocular Tumor or Melanoma |
| If you are using any medications for your eyes, please list the medications and describe how often your take them? | |

03/20/2023 3:39pm

projectredcap.org



| If you have ever had eye surgery or laser treatment related to any eye condition, please describe. | |
|---|---|
| Does anyone in your family have glaucoma? | ○ Yes ○ No ○ Maybe, Not sure |
| If YES, who has glaucoma (relationship)? | |
| ☐ Mother ☐ Father ☐ Sister ☐ Brother ☐ Daughte ☐ Grandfather ☐ Other | r □ Son □ Grandmother |
| Does anyone in your family have a history of blindness? | ○ Yes ○ No ○ Maybe, Not sure |
| If YES, who has a history of blindness (relationship)? | |
| ☐ Mother ☐ Father ☐ Sister ☐ Brother ☐ Daughte ☐ Grandfather ☐ Other | r □ Son □ Grandmother |
| END TIME for Ocular and Medical History | |
| | 8 |
| Warning: It has been over 30 minutes since the start time. Please check the start time and end time on this | Yes No<br>(The time period is over 30 minutes.) |

REDCap\* 03/20/2023 3:39pm projectredcap.org

SIGHT Page 1

# Vision Screening Snellen And IOP Results

| Record ID | |
|---|---|
| Start Time Visual Acuity | |
| | (Time CIRCLE am / pm) |
| Subject ID | |
| | (Study ID= CDC + Initials + Record ID) |
| Visual Acuity and IOP completed by | ○ UAB team ○ Self-Administered |
| Visual Acuity and IOP completed by (Name/#) | |
| | - |
| Visual Acuity (Snellen Results): Look at the Med subject wears prescription eye glasses. Ask the | |
| If the subject wears glasses, are they wearing them today f | for the visual acuity test? |
| ○ Yes (With Correction) ○ No (W/O Correction) | |
| Visual Acuity Right Eye | |
| ○ 20/20 ○ 20/25 ○ 20/30 ○ 20/40 ○ 20/50 ○ 20/200 ○ CF ○ HM ○ LP ○ NLP ○ 20/400 | |
| Visual Acuity Left Eye | |
| ○ 20/20 ○ 20/25 ○ 20/30 ○ 20/40 ○ 20/50 ○ 20/200 ○ CF ○ HM ○ LP ○ NLP ○ 20/400 | 20/60 |
| Does the subject use any low vision aids for reading, using the computer, or telephone? Read the following choices. | |
| Is the subject legally blind and requires referral for low vision | on services? |
| ○ Yes ○ No | |
| End Time for Visual Acuity | |
| | (Time CIRCLE am / pm) |
| Warning: It has been over 30 minutes since the start time. Please check the start time and end time of visual acuity. | Yes No (The time period is over 30 minutes.) |
| 03/20/2023 3:39am | projectredcap.org REDCap |

| Autorefraction Results | |
|---|---|
| Autorefraction OD | |
| Autorefraction OS | |
| | <del></del> |
| Fue Bressure (IOB) Heine I Core Tomometer | |
| Eye Pressure (IOP) Using I-Care Tomometer | |
| Start Time Eye Pressure (IOP) | |
| | (Time CIRCLE am / pm) |
| Intraocular Pressure (IOP) Right Eye (OD) | Left Eye (OS) |
| IOP measurement 1 | |
| IOP measurement 2 | |
| IOP measurement 3 | |
| 9 | |
| IOP Measurement (OD- right eye) | |
| | (range 1-60 mmHg) |
| IOP Measurement (OS-left eye) | |
| TOP Preusurement (OS-reit eye) | · |
| | (range 1-60 mmHg) |
| Since IOPs in First Reading >21, Measure Again | |
| IOP (OD-right eye): 2ND Reading | |
| | (2nd Reading Range 1-60 mmHg) |
| IOP (OS-left eye): 2ND Reading | |
| | (2nd Reading Range 1-60 mmHg) |
| The IOP Readings in 1ST and 2ND Time Differ More Than 2, Ne | eed 3RD Reading |
| IOP (OD-right eye) : 3RD Reading | |
| | (3RD Reading Range 1-60 mmHg) |
| IOP (OS-left eye): 3RD Reading | |
| tor to stere eye, sho heading | (222.2 |
| | (3RD Reading Range 1-60 mmHg) |
| Final IOP (OD-right eye) Reading: If IOP(OD) were | |
| measured 3 times, use middle value; If measured twice, use mean (average) value. | |
| Final IOP (OS-left eye) Reading: If IOP(OS) were | |
| measured 3 times, use median; If measured twice, use | - |
| mean value | |

03/20/2023 3:39pm

projectredcap.org



| RY . | |
|---|---|
| IOP greater than 30, subject requires FAST TRACK | |
| ○ Yes ○ No | |
| FAST TRACK RECOMMENDATIONS | |
| <ul> <li>○ FAST TRACK- Schedule with eye care provider within 1 Day</li> <li>○ FAST TRACK- Schedule with eye care provider within 1 W</li> <li>○ FAST TRACK- Schedule with an eye care provider within 2</li> </ul> | eek (IOP>35) |
| When is FAST TRACK subject scheduled for eye exam? | |
| | (Date and Time) |
| Where is FAST TRACK subject scheduled for eye exam? (Date and Time) | |
| <ul> <li>UAB Department of Ophthalmology</li> <li>UAB Lions Eye Clinic</li> <li>David Allgood, OD Centreville</li> <li>Own eye care provider ( get record release)</li> </ul> | |
| End Time for IOP | |
| Warning: It has been over 30 minutes since the start time. Please check the start time and end time of IOP. | Yes No (The time period is over 30 minutes.) |
| Vision Screening Failure | |
| Did subject meet any of the below criteria (Check all that ap | ply): |
| ☐ 20/40 or worse in either eye<br>☐ IOP > OR equal to 23 mmHg | |
| Name of referral doctor or practice | |

REDCap\* 03/20/2023 3:39pm projectredcap.org

# **Nei Vision Function Quesionnaire9**

| Record ID | | : |
|---|---|---|
| START TIME NEI VFQ-9 | | |
| Subject Name/Initials: | | |
| Study ID | | |
| | (Study ID= CDC + Initials + Record | ID) |
| Date NEI-VFQ | - | |
| NEI VFQ-9 completed by | ○ UAB team ○ Self-Administere | d |
| NEI-VFQ-9 completed by (Name/#) | | |
| GENERAL VISION: At the present time, would you say your lenses, if you wear them) is: | eyesight using both eyes (with glasses o | or contact |
| ○ Excellent ○ Good ○ Fair ○ Poor ○ Very poor | Completely blind | |
| 2. WELL-BEING/ MENTAL HEALTH: How much of the time do | you worry about your eyesight? | |
| <ul> <li>None of the time</li> <li>A little of the time</li> <li>Some of the time</li> <li>Most of the time</li> <li>All of the time</li> </ul> | | |
| 3. NEAR VISION, READING NORMAL NEWSPRINT: How much newspapers? Would you say you have: | difficulty do you have reading ordinary p | rint in |
| <ul> <li>No difficulty at all</li> <li>A little difficulty</li> <li>Moderate difficulty</li> <li>Extreme difficulty</li> <li>Stopped doing this because of you eyesight</li> <li>Stopped doing this for other reason or not interested in do</li> </ul> | oing this | |
| 4. NEAR VISION, SEEING WELL UP CLOSE: How much difficult see well up close, such as cooking, sewing, fixing things around the second second services. | | |
| <ul> <li>No difficulty at all</li> <li>A little difficulty</li> <li>Moderate difficulty</li> <li>Extreme difficulty</li> <li>Stopped doing this because of your eyesight</li> <li>Stopped doing this for other reasons or not interested in contract the contract of the contract of</li></ul> | doing this | |
| 03/20/2023 3:39pm | projectredcap.org | REDCap |